CLINICAL TRIAL: NCT01393847
Title: Biochemical and Genetic Mechanisms for Etiology of Sickle Cell Pain
Brief Title: Nitric Oxide and Sickle Cell Pain
Status: Terminated | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110189; 11-NR-0189
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2013-12-05

CONDITIONS: Sickle Cell Disease; Pain
Keywords: Sickle Cell; Pain; Genetics; Sickle Cell Disease; Healthy Volunteer; HV
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Sickle cell disease often causes crises, with episodes of pain. Many people with sickle cell disease also have pain between crises. Inflammation is an important part of sickle cell pain. It may be related to levels of nitric oxide. Nitric oxide is a gas in the body that helps relax blood vessels and may be related to the pain from sickle cell disease. Researchers want to study the relationship between blood levels of nitric oxide and pain in people with sickle cell disease. Researchers also want to study how certain genes express themselves related to sickle cell pain.

Objectives:

- To collect blood samples and other genetic expression information to study sickle cell pain and its relation to nitric oxide levels in the blood.

Eligibility:

* People at least 18 years of age who have sickle cell disease.
* Healthy volunteers at least 18 years of age.

Design:

* This study requires a screening visit and four study visits scheduled 1 week apart. Each visit will last about 1 hour.
* Participants will be screened with a medical history and physical exam. They will complete questionnaires about pain levels (if any). They will also provide blood samples for genetic and other testing.
* Participants will have a breath test to see how much nitric oxide they exhale. They will also have a test of their ability to detect small changes in temperature and touch.
* Participants will keep a diary to record daily pain levels and pain medicines taken. They will write down what they eat to track foods that contain nitrates (such as meats like ham and bacon and vegetables like beets and spinach).
* At each of the four study visit, participants will bring the pain diary, provide blood samples, and have breath nitric oxide tests.

DETAILED DESCRIPTION:
Sickle cell disease is a systemic disorder whose proximate cause is a mutation in the beta-globin chain of hemoglobin. Although it is characterized by differing degrees and patterns of clinical manifestations, its major features include severe episodes of pain. The sickle cell pain crisis is one of the most typical characteristics of this disease and pain associated with crisis is reported to be more intense than other types of clinical pain by those with sickle cell disease and displays both nociceptive and neuropathic qualities. Pain in sickle cell disease is more widely experienced and poorly managed than previously considered. In one community sample, more than 50 percent of the patients reported experiencing pain on more than half the days of the study period. Painful crisis consist of pain experienced in different areas of the body, typically in the extremities, back, abdomen and chest and some studies suggest that patients experience prodromal or pre-crisis phases of their pain, some of which last up to 24 hours before developing the typical features of a pain crisis. The nature of pain experience in patients with sickle cell disease is not well documented nor are the mechanisms of sickle cell pain well understood.

Objectives: The first objective of the study is to characterize genetic expression data of sickle cell disease and matched controls at weekly time points over a 4 week period. The second objective is to measure levels of exhaled Nitric Oxide (eNO) and other biomarkers in sickle cell patients and in matched controls over the same time points. The third objective is to evaluate experimental pain perception in both groups.

Population: By stratifying patients by pain level, this study will recruit sickle cell patients with a range of symptom severity (N=45) and sex-, race-, ethnicity and age-matched controls (N=45) without sickle cell trait from the NIH Patient Recruitment and Referral Service.

Design: This is a prospective, exploratory study of steady state and acute pain phase in sickle cell patients. Participants will undergo evaluations (eNO and blood collection) during weekly clinic visits and keep a pain diary for 4 weeks after the first visit. All participants will also undergo one session of quantitative sensory testing.

Importance: The purpose of this study is to improve the understanding of the biochemical and molecular genetic mechanisms associated with sickle cell pain by characterizing the transcriptome of sickle cell disease during steady state and pain phases. It is hypothesized that analysis of the transcriptome will result in a panel of biomarkers that correlate with the severity level of pain and perhaps signal the onset of a painful episode. The successful elucidation of these relationships may identify novel targets for intervention leading to attenuation of sickle cell pain, improved treatment and less impact on quality of life and functional status.

ELIGIBILITY:
* INCLUSION CRITERIA FOR SICKLE CELL SUBJECTS:

All subjects with sickle cell disease will be eligible for enrollment in this study if they meet all of the following criteria:

18 years of age or older

Diagnosis of sickle cell disease (electrophoretic or HPLC documentation of hemoglobin S only phenotype is required)

No vaso-occlusive crisis during the previous two weeks

Medically stable

Can speak and understand English to complete assessments and scales

INCLUSION CRITERIA FOR MATCHED CONTROLS:

All volunteer matched control study participants will be eligible for enrollment on this study if they meet all the following criteria:

18 years of age or older

Non-sickle cell trait or disease

Medically healthy based upon the history and physical exam and screening blood analyses

No chronic pain condition.

Can speak and understand English to complete assessments and scales

Ethnicity, age (within 5 years), and sex matched to that of sickle cell subjects already enrolled on study

EXCLUSION CRITERIA FOR ALL STUDY PARTICIPANTS:

Study participants will be excluded from the study if he/she has one or more of the following:

Inability to provide his/her own informed consent.

Drug or alcohol dependence/abuse within the past 5 years

Cigarette smoking or the use of any tobacco products within two years

Use of tranquilizers, steroids, non-steroidal anti-inflammatory agents three or more times per week.

Clinically significant medical condition that will confound the analysis of factors associated with sickle cell pain, such as:

* Chronic inflammatory disease (i.e. rheumatoid arthritis, systemic lupus erythematosus, cirrhosis)
* Diabetes mellitus
* Uncontrolled hypertension
* Known malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06-17; Study Completion 2013-12-05

PRIMARY OUTCOMES:
Difference in whole blood gene expression in the peripheral blood of sickle cell subjects and matched controls during pain and pain-free states.

SECONDARY OUTCOMES:
Quantification of pain sensory perception, eNO, and laboratory correlates in sickle cell subjects and in matched controls

CONTACTS AND LOCATIONS:
Overall Officials: Alan N Schechter, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schechter AN. Hemoglobin research and the origins of molecular medicine. Blood. 2008 Nov 15;112(10):3927-38. doi: 10.1182/blood-2008-04-078188. PMID 18988877
- [Background] Hagar W, Vichinsky E. Advances in clinical research in sickle cell disease. Br J Haematol. 2008 May;141(3):346-56. doi: 10.1111/j.1365-2141.2008.07097.x. Epub 2008 Mar 12. PMID 18341629
- [Background] McClish DK, Smith WR, Dahman BA, Levenson JL, Roberts JD, Penberthy LT, Aisiku IP, Roseff SD, Bovbjerg VE. Pain site frequency and location in sickle cell disease: the PiSCES project. Pain. 2009 Sep;145(1-2):246-51. doi: 10.1016/j.pain.2009.06.029. Epub 2009 Jul 23. PMID 19631468